CLINICAL TRIAL: NCT05286827
Title: Phase II Study of Olaparib in Subjects With Advanced Pancreatic Acinar Cell Carcinoma
Brief Title: Olaparib in Subjects With Advanced Pancreatic Acinar Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000596; 000596-C
Record Dates: First submitted 2022-03-12; First posted 2022-03-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03-31

CONDITIONS: Pancreatic Acinar Cell Carcinoma
Keywords: Poly-Adp Ribose Polymerase (Parp)-1 Inhibitor; Homologous Recombination Repair; Platinum-Sensitive
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Olaparib, taken orally, twice daily
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Administered orally (300 mg) twice daily continuously for 28-day cycles for up to 2 years.

SUMMARY:
Background:

Pancreatic Acinar Cell Carcinoma (PACC) is a rare pancreatic tumor. People with PACC usually present with advanced disease, and their prognosis is poor. Researchers want to learn if a cancer drug called olaparib can help.

Objective:

To see if olaparib is an effective treatment for PACC.

Eligibility:

People aged 18 and older with PACC whose cancer did not respond to previous treatments or is not eligible for surgery.

Design:

Participants will be screened with the following:

Medical history

Physical exam

Blood and urine tests

Electrocardiogram (to test heart function)

Computed tomography (CT) scans

Pregnancy test (if needed)

Tumor biopsy (if a sample is not available)

Treatment will be given in 28-day cycles. Participants will take olaparib by mouth twice daily for each cycle. They will keep a medicine diary. They will receive treatment for up to 2 years. They may stop treatment early if their cancer gets worse or they have serious side effects.

Participants will have study visits at the beginning of each cycle. At visits, they will repeat some screening tests. They will be asked about any changes in medicines they are taking and how they are feeling. They will have CT scans every 8 weeks starting in cycle 2.

Participants will give blood samples for research. They may have optional tumor biopsies.

Participants will have 2 follow-up visits in the 30 days after treatment ends or before they begin a new anti-cancer treatment. Then they will be contacted every 3 months by phone for 1 year.

Participation will last for up to 3 years.

DETAILED DESCRIPTION:
Background:

* Pancreatic Acinar Cell Carcinoma (PACC) is a rare pancreatic tumor, representing 0.5-1% of all pancreatic malignancies.
* PACC is commonly advanced at presentation and median overall survival in this population is poor.
* PACC is pathologically and biochemically distinct from pancreatic adenocarcinoma.
* No clinical trials for PACC have ever been reported.
* Patients are most commonly treated with combination regimens used for either pancreatic or colon adenocarcinoma with poor (approximately 30%) response rates in the first-line setting.
* PACC pathological specimens demonstrate evidence of high chromosomal instability, a hallmark of DNA repair deficiency.
* Data derived from ovarian and prostate cancer patients has demonstrated that mutations in DNA repair genes can define subgroups of cancer patients with distinct vulnerabilities to DNA damage response inhibitors.
* Olaparib is a Poly-ADP ribose polymerase (PARP)-1 inhibitor that has been FDA approved for the treatment of BRCA-mutant homologous recombination repair (HRR) deficient cancers.
* As PACC has multiple hallmarks of HRR deficiency, we hypothesize that PACC will be sensitive to PARP inhibition with olaparib.
* Pre-clinical modeling of PACC has been very limited with no currently available animal models or cell lines, which precludes testing this hypothesis in the laboratory setting.

Objective:

- To assess the anti-tumor activity of single agent olaparib, a PARP inhibitor, in participants with advanced pancreatic acinar cell carcinoma (PACC)

Eligibility:

* Participants must have advanced previously treated PACC
* Age >=18 years
* Adequate organ and bone marrow function

Design:

* This is a phase II, single arm, single center study of olaparib in participants with advanced previously treated PACC.
* All participants will take olaparib by mouth twice daily for up to two years or until disease progression or intolerable side effects.
* Participants will be assessed for safety (continuously) and efficacy (every 8 weeks).
* Up to 13 evaluable participants will be enrolled.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Histological or cytological diagnosis of pancreatic acinar cell carcinoma (PACC) as confirmed by NIH Laboratory of Pathology (LP).
2. Participants must have received one prior line of combination chemotherapy (or be ineligible to receive combination chemotherapy) with tumor still not amenable for potentially curative resection or be ineligible to receive combination chemotherapy. There is no limit on the number of prior therapies.
3. Access to medical records from past treatment
4. Measurable disease, per RECIST 1.1.
5. Age >=18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status <=1.
7. At least 3 weeks from previous chemotherapy or radiation therapy prior to planned start of treatment.
8. At least 30 days or 5 half-lives (whichever is greater) since receipt of any investigational therapy prior to planned start of treatment.
9. Fully recovered from all reversible sequalae and >=2 weeks from major surgery or from minor surgical procedure such as biliary or duodenal stenting prior to planned start of treatment.
10. At least 2 weeks since last use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil).
11. At least 5 weeks since last use of phenobarbital, enzalutamide, and at least 3 weeks since last use of other strong (e.g., phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John s Wort) or moderate (e.g., bosentan, efavirenz, modafinil) CYP3A inducers.
12. Adequate organ and marrow function as measured within 28 days prior to study treatment as defined below:

    * leukocytes >=3,000/mcL
    * absolute neutrophil count >=1,500/mcL
    * hemoglobin >= 10 g/dL with no blood transfusion within the last 28 days
    * platelets >=100,000/mcL
    * total bilirubin within 1.5x normal institutional upper limit of normal (ULN)
    * Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) <= institutional ULN unless liver metastases are present in which case they may be <=5x ULN
    * Creatinine must be within normal range, OR >=51 mL/min per the formula below* or measured by 24-hour urine test

      * Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F) serum/ creatinine (mg/dL) x 72^a, where F=0.85 for females and F=1 for males

    This list includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.
13. The effects of olaparib on the developing human fetus are unknown. For this reason and because PARP inhibitor agents are known to be teratogenic, individuals of child-bearing potential (IOCBP) and individual able to father a child must agree to use adequate contraception prior to study entry and for the duration of study participation.
14. Participants must agree to abstain from consuming grapefruit juice throughout the duration of study treatment with olaparib.
15. Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib.
2. Participants unable to swallow orally administered medication or suffering from gastrointestinal (GI) disorders likely to interfere with absorption of study medication.
3. Participants with human immunodeficiency virus (HIV) are excluded even if viral load is undetectable
4. Active hepatitis B (HBV) or hepatitis C virus (HCV)
5. Resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or participants with congenital long QT syndrome.
6. Recent (within 3 months) myocardial infarction
7. Unstable angina pectoris.
8. Symptomatic congestive heart failure
9. Uncontrolled major seizure disorder
10. Superior vena cava syndrome
11. Extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan
12. Psychiatric illness/social situations (within the last 3 months) that would limit compliance with study requirements or prohibits obtaining informed consent
13. Uncontrolled intercurrent illness or participants considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active uncontrolled infection as documented in prior records or suggested by medical history, physical examination or standard clinical assessments such as imaging and laboratory studies
14. Myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
15. Solid or liquid malignancy other than PACC unless curatively treated with no evidence of disease for >=5 years, except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.
16. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
17. Participants who are nursing and unwilling to stop.
18. Symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. Brain metastases are considered uncontrolled if the dose of corticosteroid being provided for control of brain metastases has been titrated in the 4 weeks prior to start of treatment.
19. Participants with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for >=28 days. Participants with unstable spinal cord compression are ineligible even if previously treated.
20. Participants with large volume ascites, serum albumin < 2.5 mg/dL, or having received paracentesis within the last 4 weeks
21. Participants with persistent toxicities > Grade 2 or with new Grade 2 events within the last 2 weeks per Common Terminology Criteria for Adverse Event (CTCAE) version 5 caused by previous cancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
antitumor activity | 1 year post-last dose of olaparib
  Objective response rate (ORR, CR+PR)

SECONDARY OUTCOMES:
anti-tumor efficacy | 1 year after last olaparib treatment
  Disease control rate, median duration of treatment response, median progression-free survival (PFS) and median overall survival (OS)
safety | from start of treatment to 30 days after last treatment
  AEs and SAEs of olaparib

CONTACTS AND LOCATIONS:
Overall Officials: Christine C Alewine, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. @@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000596-C.html